CLINICAL TRIAL: NCT05400291
Title: Gag-layer in the Urothelium of the Human Upper Urinary Tract
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Ferring Ventures (Unknown)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor. MD, Aarhus University Hospital
Other Study IDs: GAG
Record Dates: First submitted 2022-02-21; First posted 2022-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer; Renal Cancer
Keywords: glykosaminoglycan layer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — a 1x1cm biopsi from the bladder or the renal pelvis along with a 1x1cm biopsi from the urether.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal Cell Carcinoma: patients undergoing radical nephrectomy because of renal clear cell carcinoma, tissue will be collected after the organ is removed.
  Interventions: Diagnostic Test: Chondroitin Sulfate Staining
- Muscle Invasive Bladder Cancer: patients underoing radical cystectomi because of muscle-invasive bladder cancer, tissue will be collected after the organ is removed.
  Interventions: Diagnostic Test: Chondroitin Sulfate Staining

INTERVENTIONS:
Diagnostic Test: Chondroitin Sulfate Staining — Staining of histopathological slides

SUMMARY:
Urothelial carcinomas of the lower and upper urinary tract can be considered "twin diseases". Much of the current clinical decision-making surrounding Upper Tract Urothelial Carcinoma (UTUC) is extrapolated from evidence that is based on urothelial carcinoma of bladder patients.

The inner wall of the bladder is coated with a substance called glycosaminoglycan (GAG). GAG is known to form a gel-like layer on the apical cell membrane and act as a barrier against urine and pathogens in the lower urinary tract.

Currently no published research on the presence of a GAG layer in the upper urinary tract exists. However, literature suggests that the ureteral utothelium can be transduced without enhancers, and the ureteral urothelium may be intrinsically different from bladder, both by the presence or absence of a GAG-layer, by different composition/thickness of the GAG-layer.

Any functional differences between the urothelial layers in the bladder and in the upper urinary tract may affect the adeno-virus transduction, which again will have potential impact on future treatment of UTUC patients with a current unmet medical need.

DETAILED DESCRIPTION:
This study will include patients either undergoing radical nephrectomy or radical cystectomy. After organ removal during surgery a biopsi (1x1 cm) will be collected from the ureter and the renal pelvis or from the ureter and the bladder (depending on type of surgery).

These biopsies will be examined and compared, using molecular biotechniques, for the presence of glykosamino glykan (GAG) layer.

There is no project related follow up for patients included, other than what is standard post-operative regime in the department.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer or renal cell carcinoma
* Ability to understand and sign informed consent form

Exclusion Criteria:

* Previous history of cancer
* Immune suppressing medication
* Treatment with local or systemic steroids (< 3 months prior to enrollment)
* Treatment with antibiotics due to urinary tract infection or pyelonephritis (< 3 months prior to enrollment)
* Previous radiation therapy of the pelvic floor
* Ureteric stent
* Dilatation of the upper urinary tract detected on imaging
* Dilatation of the upper urinary tract detected on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cystectomy or nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of a GAG layer in the upper urinary tract | samples are collected and stained immediately after the surgery, all samples will be compared and analyzed once all samples have been collected
  Number of specimens with presence of GAG layer by histopatological staining

SECONDARY OUTCOMES:
Thickness of the potential GAG layer in the upper urinary tract | samples are collected and stained immediately after the surgery, all samples will be compared and analyzed once all samples have been collected
  Compare the morphological and histological features of a GAG layer in the upper urinary tract to that of the bladder

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B Jensen, Dr. Med., Principal Investigator — AUH
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark